CLINICAL TRIAL: NCT00338481
Title: "Red Morphine Drops" for Symptomatic Treatment of Dyspnoea in Terminal Patients With Primary Lung Cancer or Lung metastases-a Pilot Study
Brief Title: "Red Morphine Drops" for Symptomatic Treatment of Dyspnoea in Lung Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sankt Lukas Hospice (Other)
Responsible Party: Torben Krantz, Sankt Lukas Hospice
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2005-060-version1a
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-02

CONDITIONS: Dyspnea; Lung Neoplasms
MeSH Terms: conditions — Dyspnea; Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Morphine p.o.
- 2 (Active Comparator)
  Interventions: Drug: Morphine s.c.

INTERVENTIONS:
Drug: Morphine p.o. — Morphine p.o. in "red morphine drops" calculated as 1/12 of the 24 hours opioid consumption converted to morphine p.o., max. 24 mg morphine p.o.and isotonic sodium chloride s.c.
  Arms: 1
Drug: Morphine s.c. — False "red morphine drops" without morphine p.o. and 60% of 1/12 of the 24 hours opioid consumption converted to morphine p.o. but given s.c., max. 14,4 mg
  Arms: 2

SUMMARY:
The purpose of this study is to test whether "red morphine drops" applied in the mouth are superior to an equivalent amount of morphine applied as subcutaneous injection for the relief of breathlessness in terminal patients suffering from primary lung cancer or lung metastases.

DETAILED DESCRIPTION:
Breathlessness or dyspnea in terminal cancer patients with lung cancer is common and opioids such as morphine is the mainstay of symptomatic treatment. Subcutaneous administration of morphine provides fast symptomatic relief, but it has been the impression in our institution that "red morphine drops" applied orally may have equal or better efficacy and faster onset time.

Comparison: Patients with lung cancer or lung metastases with moderate to severe dyspnea at rest are treated with either orally applied "red morphine drops" or an equivalent amount of morphine applied subcutaneously.

ELIGIBILITY:
Inclusion Criteria:

* Primary lung cancer or lung metastases and
* Moderate to severe dyspnea at rest (VAS equal to or more than 30)

Exclusion Criteria:

* Causal treatment of dyspnea possible and indicated
* Not receiving opioids on a regular basis
* Methadone treatment
* Intolerance to morphine
* Without understanding of patient information
* Depressed consciousness
* Oxygen treatment, if changed with-in 20 min before start
* Short-acting opioids with-in 4 h before start
* Inhalation therapy for bronchodilation with-in 20 min before start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Dyspnea on a VAS scale | 1 hour

SECONDARY OUTCOMES:
Respiratory rate, pulse rate, oxygen saturation | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Torben Krantz, Physician, Principal Investigator — Sankt Lukas Hospice
Locations (1):
- Sankt Lukas Hospice, Copenhagen, Hellerup, Denmark